CLINICAL TRIAL: NCT01973881
Title: Quantitative MRI for Myelofibrosis - MRI Parameters as Biomarkers for Analyzing Extent of Disease and Measuring Response to Treatment
Brief Title: Quantitative MRI for Myelofibrosis
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Sanofi (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UMCC 2014.034; R01CA238023 (NIH); HUM00077505 (Other: University of Michigan)
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- T1 weighted MRI (magnetic resonance imaging): For the development and validation of functional magnetic resonance imaging (MRI) parameters as biomarkers for analyzing extent of disease and quantifying response to treatment in patients with myelofibrosis. Quantitative MRI parameters for diffusion of water and/or fat content in bone marrow will determine extent of disease in patients with myelofibrosis, and changes in these parameters will predict response to therapy. To investigate this hypothesis, the researchers will perform this pilot clinical study of diffusion and fat content (T1 weighted imaging) in patients before and during treatment for myelofibrosis. The researchers expect to identify MRI parameters that determine the extent and severity of bone marrow disease in these patients and determine response to therapy at earlier time points than currently used clinical parameters.
  Interventions: Procedure: T1 Weighted MRI (magnetic resonance imaging)

INTERVENTIONS:
Procedure: T1 Weighted MRI (magnetic resonance imaging) — Enrolled subjects will have an MRI scan performed at baseline (within 1 month before beginning therapy), at the time of a scheduled bone marrow biopsy or end of treatment cycle (6 months), and after 12 months.
  Please note: Patients in this study will be treated with chemotherapy as determined by the hematologist or the treatment protocol for an independent clinical trial for therapy of myelofibrosis. Treatment and monitoring will be performed under the usual standard of care that includes physical examinations, laboratory testing, and other indicated imaging examinations.

SUMMARY:
This study is for the development and validation of functional magnetic resonance imaging (MRI) parameters as biomarkers for analyzing extent of disease and quantifying response to treatment in patients with myelofibrosis.

DETAILED DESCRIPTION:
This study is for the development and validation of functional magnetic resonance imaging (MRI) parameters as biomarkers for analyzing extent of disease and quantifying response to treatment in patients with myelofibrosis. Quantitative MRI parameters for diffusion of water and/or fat content in bone marrow will determine extent of disease in patients with myelofibrosis, and changes in these parameters will predict response to therapy. To investigate this hypothesis, the researchers will perform this pilot clinical study of diffusion and fat content (T1 weighted imaging) in patients before and during treatment for myelofibrosis. The researchers expect to identify MRI parameters that determine the extent and severity of bone marrow disease in these patients and determine response to therapy at earlier time points than currently used clinical parameters. This research will lay the foundation for larger clinical trials using MRI to assess and predict effects of existing and new therapeutic agents for patients with myelofibrosis.

This study proposes that more advanced MRI techniques currently used in clinical medicine can be applied to enable response to therapy to be determined earlier than currently is possible for patients with myelofibrosis. In particular, this study is designed to determine to what extent abnormalities in diffusion of water molecules (diffusion MRI) and/or fat content in bone marrow (T1-weighted imaging) define extent of initial disease and serve as early predictors of response to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male /female subjects over the age of 18
2. Diagnosis of primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocythemia myelofibrosis.
3. No contraindications to MRI
4. Able to undergo MRI without anesthesia

   -

Exclusion Criteria:

1. Patients with pacemakers or other implanted magnetic devices that may malfunction or move because of the strong magnetic field inside the MRI room and scanner.
2. Any prior adverse event associated with MRI that is not related to injection of contrast agents or other medicines.

   -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People diagnosed with myelofibrosis who are able to undergo an MRI without anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2014-12-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Using MRI to assess treatment response in subjects with myelofibrosis | 5 years
  For the development and validation of functional magnetic resonance imaging parameters as biomarkers for analyzing extent of disease and quantifying response to treatment in patients with myelofibrosis. Quantitative MRI parameters for diffusion of water and/or fat content in bone marrow will determine extent of disease in patients with myelofibrosis, and changes in these parameters will predict response to therapy. To investigate this hypothesis, the researchers will perform this pilot clinical study of diffusion and fat content (T1 weighted imaging) in patients before and during treatment for myelofibrosis. The researchers expect to identify MRI parameters that determine the extent and severity of bone marrow disease in these patients and determine response to therapy at earlier time points than currently used clinical parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Luker, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robison TH, Levinson A, Lee W, Pettit K, Malyarenko D, Kandarpa M, Johnson TD, Chenevert TL, Ross BD, Talpaz M, Luker GD. Quantitative MRI Assessment of Bone Marrow Disease in Myelofibrosis: A Prospective Study. Radiol Imaging Cancer. 2025 Nov;7(6):e240501. doi: 10.1148/rycan.240501. PMID 41236389